CLINICAL TRIAL: NCT06913595
Title: Extended Venous Thromboemboism Prophylaxis After Bariatric Surgeries: A Comparison Of Low Molecular Weight Heparin With Direct Oral Anticoagulant
Brief Title: Low Molecular Weight Heparin vs Direct Oral Anticoagulant After Bariatric Surgery
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Elshwadfy Nageeb, lecturer of general surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N-55-2024
Record Dates: First submitted 2025-03-24; First posted 2025-04-06 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Deep Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — N(4)-oleylcytosine arabinoside; Enoxaparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Molecular Weight Heparin (Active Comparator): Low molecular weight heparin as aprophylaxis after bariatric surgery
  Interventions: Drug: Low Molecular Weight Heparine
- Direct Oral Anticoagulant. (Experimental): Direct Oral Anticoagulant as aprophylaxis after bariatric surgery
  Interventions: Drug: Direct Oral Anticoagulant.

INTERVENTIONS:
Drug: Direct Oral Anticoagulant. — Direct Oral Anticoagulant AFTER BARIATRIC SURGERY
  Other Names: RIVROXABAN
  Arms: Direct Oral Anticoagulant.
Drug: Low Molecular Weight Heparine — Low molecular weight heparin after bariatric surgery
  Other Names: Enoxaparine
  Arms: Low Molecular Weight Heparin

SUMMARY:
Extended Venous Thromboemboism Prophylaxis After Bariatric Surgeries: A Comparison Of Low Molecular Weight Heparin With Direct Oral Anticoagulant

DETAILED DESCRIPTION:
This study aims to compare the effectiveness of rivaroxaban versus low molecular weight heparin in reducing the incidence of PMVT after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

- BARIATRIC PATIENTS

Exclusion Criteria:

* BLEEDING TENDENCY

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-10-25 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
VENOUS THROMBOEMBOLISM | 1 year
  DVT after bariatric surgery

CONTACTS AND LOCATIONS:
Overall Officials: mohammed elshwadfy, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No